CLINICAL TRIAL: NCT06846359
Title: The Impact Of Gastric Phenotyping In Predicting And Assessing The Clinical Success Of Gut-Directed Hypnotherapy For Patients With Gastroduodenal DGBIS.
Brief Title: Treatment of Upper Gastrointestinal Symptoms Using Hypnotherapy Sessions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiao Jing (Iris) Wang, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-007628
Record Dates: First submitted 2025-02-12; First posted 2025-02-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: GI Symptoms
Keywords: hypnotherapy; disorders of gut-brain interaction
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hypnotherapy (Experimental): 7 pre-recorded hypnotherapy sessions delivered over 12 weeks via patient's own electronic device. Sessions are approximately 40 minutes long.
  Interventions: Behavioral: Hypnotherapy
- Educational module (Other): Patient's will be given a link to a educational module that reviews chronic GI conditions, pathophysiology, and alternative treatment options.
  Interventions: Behavioral: Educational module

INTERVENTIONS:
Behavioral: Hypnotherapy — Seven pre-recorded hypnotherapy sessions delivered over the course of twelve weeks via the patient's own electronic device such as a smartphone, tablet, or laptop. The length of the audio-recorded treatment sessions is expected to be approximately 40 minutes on average.
  Arms: Hypnotherapy
Behavioral: Educational module — self-guided online module reviewing chronic GI conditions, pathophysiology, and alternative treatment options.
  Arms: Educational module

SUMMARY:
The purpose of this research is to evaluate if hypnotherapy delivered digitally will help your GI symptoms.

DETAILED DESCRIPTION:
This study will assess the effects of digitally delivered hypnotherapy sessions n those with upper GI symptoms. There are 2 therapy arms: Hypnotherapy treatment over 3 months or control arm with an educational module. The hypnotherapy treatment consists of seven pre-recorded hypnotherapy sessions that will be digitally delivered to patients on their own electronic devices via an existing digital platform provided by metaMe Health. metaMe Health is a company specialized in the delivery of digital hypnotherapy protocols. The sessions will be delivered to patients over twelve weeks in accordance with current gut-direct hypnotherapy practice. The patients must agree to have their consent and content delivered electronically and provide periodic outcomes by completing electronic symptom questionnaires. Both arms will also complete C13 breath test and gastric alimetry testing before and after being randomized.

The whole study will last for 24 weeks: the initial 12-week treatment period and then an additional 12-week follow-up period

ELIGIBILITY:
Inclusion criteria:

* Patients will meet criteria for at least one upper GI DGBI including functional dyspepsia, any nausea/vomiting disorder, or functional abdominal bloating. Lower GI DGBIs, such as IBS, are allowable if the primary symptom is either an upper GI symptom or bloating/distension.
* Participants will have had a negative 4-hour solid food gastric emptying test previously or a normal C13 Breath test at screening.
* Patients with known disaccharide intolerances may be included if dietary restrictions are maintained during the duration of the study.
* Patients utilizing cannabinoid based substances may be included if no dose changes are made during the duration of the study
* Patients will be proficient in English language for comprehension of content
* Patients will have reliable access to digital delivery systems for content and questionnaire access via smartphone over the course of the study and follow up period.

Exclusion criteria:

* Patients with known current diagnosis of small intestinal bacterial overgrowth (SIBO), gastroparesis, rumination syndrome, chronic intestinal pseudo-obstruction, advanced connective tissue diseases (e.g. scleroderma), and uncontrolled inflammatory bowel disease (IBD) will be excluded.
* Patients with current untreated H. pylori infection will be excluded.
* In patients with predominant bloating symptoms and constipation, those with untreated pelvic floor dysfunction will be excluded. If the predominant symptoms are nausea/vomiting or dyspepsia, or if constipation is not present, then pelvic floor dysfunction will not be exclusionary.
* Patients who have a history of cognitive delay, traumatic brain injury with residual deficits, history of cerebral vascular accident with residual deficiencies in cognition, dementia, shall be excluded
* Patients with significant psychiatric illness with component of psychosis (schizophrenia, bipolar disorder), as well as severe untreated major depressive disorder with suicidal ideation will be excluded
* Patients with substance abuse disorders and drug addiction will be excluded.
* Patients who are unlikely to comply or unlikely to benefit from psychotherapy-based interventions may be excluded at the direction of medical screening provider or principal investigator.
* Standard inclusion criteria will include: ability to provide informed consent, absence of other diseases (structural or metabolic) which could interfere with interpretation of the study results.
* Stable doses medications are permissible, but dosing should not be changed during study period.
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Irritable Bowel Symptom Severity Index (IBS-SSS) score | Baseline, 12 weeks, 24 weeks
  The Irritable Bowel Syndrome Symptom Severity Scale (IBS-SSS) is a 5-item questionnaire that rates the severity of abdominal pain, number of days with abdominal pain, distention/bloating, bowel habits, and interference in quality of life. Each question has a possible score of 100 points. The total score can range from 0 - 500, with higher scores indicating greater severity of symptoms.
Change in Patient Assessment of Upper Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) score | Baseline, 12 weeks, 24 weeks
  The Patient Assessment of Upper Gastrointestinal Disorders Symptom Severity Index (PAGI-SYM) is a 20-item questionnaire that rates the severity of upper gastrointestinal symptoms across 6 subscales: heartburn, nausea/vomiting, fullness, bloating, upper abdominal pain, and lower abdominal pain. Subscale scores are calculated by averaging across items comprising the subscale; scores vary from 0 (none or absent) to 5 (very severe).

SECONDARY OUTCOMES:
Change in Gastroparesis Cardinal Symptom Index (GCSI) score | Baseline, 12 weeks, 24 weeks
  The Gastroparesis Cardinal Symptom Index (GCSI) is a 9-item questionnaire that assesses the severity of nine gastroparesis symptoms, grouped into three categories: nausea/vomiting, bloating, and postprandial fullness. Each symptom is rated on a scale of 0 (no symptom) to 5 (very severe). The GCSI score is calculated as an average for each category, with higher numbers indicating a greater severity of symptoms.
Change in abdominal girth | Baseline, 12 weeks
Change in Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) | Baseline, 12 weeks, 24 weeks
  The Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) is a 30-item questionnaire that assesses the quality of life for patients with upper gastrointestinal disorders. Symptom severity is rated on a 6-pointLikert scale with 0 = 'None of the time' and 6 = 'All of the time'. Higher scores indicate a poorer quality of life.
Change in Personal Health Questionnaire Depression Scale (PHQ-8) | Baseline, 12 weeks, 24 weeks
  The Personal Health Questionnaire Depression Scale (PHQ-8) is an 8-item questionnaire used to assess symptoms of depression over the last 2 weeks. Questions are rated on a 4-point Likert scale with 0 = 'Not at all sure' and 4 = 'Nearly every day'. Total scores range from 0-24, with 0-4: No significant depressive symptoms, 5-9: Mild depression, 10-14: Moderate depression, 15-19: Moderately severe depression, and 20-24: Severe depression.
Change in Work Productivity and Activity Impairment - General Health (WPAI-GH) | baseline, 12 weeks, 24 weeks
  The Work Productivity and Activity Impairment - General Health (WPAI-GH) Questionnaire is a 6-item instrument to measure impairments over the past 7 days in both paid work and unpaid work due to one's health.
Patient history files will be audited and included into the analysis to look for contributing clinical information for the development of a clinical decision rule. | End of study analysis, roughly 1 year
Satisfaction with digital delivery platform will be assessed utilizing survey at the end of treatment. | 12 weeks
Change in EQ-5D | Baseline, 12 weeks, 24 weeks
  The EQ-5D (not an abbreviation) is a 5-item questionnaire used to assess quality of life over 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Questions are rated on a 5-point Likert scale where 0 indicates no interference with daily activities, and 5 indicates inability to perform daily tasks. Higher overall scores indicate a greater degree of difficulty performing daily tasks.
Change in General Anxiety Disorder 7-item (GAD 7) | Baseline, 12 weeks, 24 weeks
  The General Anxiety Disorder 7-item (GAD 7) scale to assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety.
Change in Perceived Stress Scale (PSS-4) | Baseline, 12 weeks, 24 weeks
  The 4-item Perceived Stress Scale (PSS) measures global perceived stress experienced by the participant over the preceding 30 days. The questions in this assessment tool ask how often the participant felt or thought a certain way during the past month. Possible answers include: 0 - never; 1 - almost never; 2 - sometimes; 3 - fairly often, and 4 - very often. Possible scores range from 0 to 20, with lower scores indicating a better outcome (less stress).
Change in Alimetry Gut-Brain Wellbeing Survey (AGBW) | Baseline, 12 weeks, 24 weeks
  The Alimetry Gut-Brain Wellbeing Survey (AGBW) is a 10-item questionnaire used to assess mental wellbeing in patients with chronic gastroduodenal symptoms. Questions are rated on a 5-point Likert scale, with 0 = 'None of the time' and 5 = 'All of the time'. Higher overall score indicates a greater impact of the patient's gastroduodenal symptoms on their mental wellbeing.
Change in Brief Illness Perception Questionnaire (BIPQ-R) | Baseline, 12 weeks, 24 weeks
  The Brief Illness Perception Questionnaire (BIPQ-R) consists of nine items rated on a scale from 0 (minimum) to 10 (maximum). The first five assess cognitive perceptions such as effect on life (item 1); duration of illness (item 2); control over illness (item 3); beliefs about the effectiveness of treatment (item 4); and experience of symptoms (item 5). Items 6 and 8 assess emotional aspects to include concern about illness and a multifaceted question about mood. Item 7 assesses degree of understanding of the illness. The final item is open-ended, asking respondents to rank the three most important factors causing their illness.
Change in Visceral Sensitivity Index (VSI) | Baseline, 12 weeks, 24 weeks
  The Visceral Sensitivity Index (VSI) is a 15-item questionnaire used to assess gastrointestinal-specific anxiety. Questions are rated on a 6-point Likert scale, with 0 = 'Strongly Agree' and 6 = 'Strongly Disagree'. Higher score overall indicates a greater degree of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Jing (Iris) Wang, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No